CLINICAL TRIAL: NCT04527107
Title: A Phase 2, Randomised, Multicentre Study to Assess the Dose Level of Multiple THR-149 Injections and to Evaluate the Efficacy and Safety of THR-149 Versus Aflibercept for the Treatment of Diabetic Macular Oedema (DME)
Brief Title: A Study to Evaluate THR-149 Treatment for Diabetic Macular Oedema
Acronym: KALAHARI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxurion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-149-002; 2019-001506-17 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- THR-149 dose level 1 (Experimental)
  Interventions: Drug: THR-149 dose level 1
- THR-149 dose level 2 (Experimental)
  Interventions: Drug: THR-149 dose level 2
- THR-149 dose level 3 (Experimental)
  Interventions: Drug: THR-149 dose level 3
- THR-149 + sham (Experimental)
  Interventions: Drug: THR-149 0.13mg
- THR-149 + aflibercept flip-over (Experimental)
  Interventions: Drug: THR-149 0.13mg + aflibercept 2mg
- Aflibercept + THR-149 flip-over (Active Comparator)
  Interventions: Drug: aflibercept 2mg + THR-149 0.13mg
- Aflibercept + sham (Active Comparator)
  Interventions: Drug: Aflibercept 2mg

INTERVENTIONS:
Drug: THR-149 dose level 1 — 3 intravitreal injections of THR-149 dose level 1, 1 month apart
  Arms: THR-149 dose level 1
Drug: THR-149 dose level 2 — 3 intravitreal injections of THR-149 dose level 2, 1 month apart
  Arms: THR-149 dose level 2
Drug: THR-149 dose level 3 — 3 intravitreal injections of THR-149 dose level 3, 1 month apart
  Arms: THR-149 dose level 3
Drug: THR-149 0.13mg — 3 intravitreal injections of THR-149 0.13mg (selected dose level), 1 month apart, followed after 1 month by a sham (pretend) injection
  Arms: THR-149 + sham
Drug: THR-149 0.13mg + aflibercept 2mg — 3 intravitreal injections of THR-149 0.13mg (selected dose level), 1 month apart, followed after 1 month by an intravitreal injection of aflibercept 2mg
  Arms: THR-149 + aflibercept flip-over
Drug: aflibercept 2mg + THR-149 0.13mg — 3 intravitreal injections of aflibercept 2mg, 1 month apart, followed after 1 month by an intravitreal injection of THR-149 0.13mg (selected dose level)
  Arms: Aflibercept + THR-149 flip-over
Drug: Aflibercept 2mg — 3 intravitreal injections of aflibercept 2mg, 1 month apart, followed after 1 month by a sham (pretend) injection
  Arms: Aflibercept + sham

SUMMARY:
Part A of the study is conducted to select the THR-149 dose level.

Part B of the study is conducted to assess the efficacy and safety of the selected dose level compared to aflibercept, up to Month 3. As from Month 3, in about half of the subjects, the effect of a single flip-over injection (aflibercept or THR-149) will be evaluated when administered 1 month after the 3 monthly injections of THR-149 or aflibercept. In the other subjects, the durability of 3 monthly injections of THR 149 or aflibercept will be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent obtained from the subject prior to screening procedures
* Male or female aged 18 years or older at the time of signing the informed consent
* Type 1 or type 2 diabetes
* BCVA ETDRS letter score ≤ 73 and ≥ 39 in the study eye (for subjects in Part A); BCVA ETDRS letter score ≤ 73 and ≥ 24 in the study eye (for subjects in Part B)
* Central involved DME (CI-DME) with CST of ≥ 320µm in men or ≥ 305µm in women, on spectral domain optical coherence tomography (SD-OCT), in the study eye
* Received ≥ 5 anti-vascular endothelial growth factor (anti-VEGF) injections for the treatment of CI-DME
* BCVA ETDRS letter score ≥ 34 in the fellow eye

Key Exclusion Criteria:

* Macular edema due to causes other than DME in the study eye
* Concurrent disease in the study eye, other than central-involved DME, that could require medical or surgical intervention during the study period or could confound interpretation of the results
* Any condition that could confound the ability to detect the efficacy of the investigational medicinal product
* Previous confounding medications / interventions, or their planned administration
* Presence of neovascularisation at the disc in the study eye
* Presence of iris neovascularisation in the study eye
* Uncontrolled glaucoma in the study eye
* Any active or suspected ocular or periocular infection, or active intraocular inflammation, in either eye
* Untreated Diabetes Mellitus
* Glycated haemoglobin A (HbA1c) > 12%
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) ETDRS letter score from Baseline, in subjects in Part B of the study | At Month 3

SECONDARY OUTCOMES:
Mean change in BCVA ETDRS letter score from Baseline, by study visit | Up to Month 6
Mean change in central subfield thickness (CST) from Baseline, by study visit | Up to Month 6
Incidence of systemic and ocular adverse events (AEs) and serious adverse events (SAEs) | Up to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — Oxurion
Locations (78):
- United States (41):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Associates, Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Salehi Retina Institute Inc., Huntington Beach, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - California Retina Consultants, Oxnard, California
  - Retina Consultants San Diego, Poway, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Retina Consultants of Southern Colorado, P.C., Colorado Springs, Colorado
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - MedEye Associates, South Miami, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sierra Eye Associates, Reno, Nevada
  - Retina-Vitreous Surgeons of Central New York, PC, Liverpool, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Retina Associates of Cleveland, Inc, Cleveland, Ohio
  - Sterling Vision, P.C. dba Oregon Retina, Eugene, Oregon
  - Tenneesse Retina, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of South Texas, P.A., San Antonio, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Macula & Retina Center, Norfolk, Virginia
  - WVU Eye Institute, Morgantown, West Virginia
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- France (6):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU de Dijon, Dijon
  - Hôpital de la Croix Rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - Fondation Rothschild, Paris
  - Hôpital Lariboisière, Paris
- Germany (6):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Internationale Innovative Ophthalmochirurgie, Düsseldorf
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Regensburg, Regensburg
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Fondazione G.B. Bietti, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Fakultná nemocnica s poliklinikou Žilina, Žilina, Slovakia
- Spain (12):
  - Hospital de la Esperanza, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital Dos de Maig, Barcelona
  - Instituto Clínico Quirúrgico de Oftalmología, Bilbao
  - METAVISIÓN ARRUZAFA, S.L.Clínica de Oftalmología de Córdoba S.L. (Hospital La Arruzafa), Córdoba
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Instituto Oftalmológico Gómez-Ulla, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Fundación de Oftalmología Médica de la Comunitat Valenciana, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (8):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Kent and Canterbury Hospital, Canterbury
  - Frimley Health NHS Foundation Trust, Frimley
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - London North West University Healthcare NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland
  - Mid and South Essex NHS Foundation Trust, Westcliff-on-Sea